CLINICAL TRIAL: NCT06390488
Title: Transcutaneous Medial Plantar Nerve Stimulation in Women With Idiopathic Overactive Bladder: A Prospective Randomized Double-blind Placebo Controlled Trial
Brief Title: Transcutaneous Medial Plantar Nerve Stimulation in Women With Idiopathic Overactive Bladder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Necmettin Yildiz, Professor Doctor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PamukkaleU.ftr-NYıldız-2
Record Dates: First submitted 2024-04-01; First posted 2024-04-30 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Urinary Bladder, Overactive
Keywords: Idiopathic overactive bladder; Transcutaneous medial plantar nerve stimulation; Urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-MPNS (Experimental): In this study, the stimulation device will be connected to the patient via channel 1, and active stimulation will be performed. Channel 2 will not be connected to the patient, thus no stimulation will be given through this channel. Both channels will utilize a stimulation protocol set to continuous mode with a frequency of 20 Hz and a pulse width of 200 ms. The intensity of the current for channel 1 (ranging from 0 to 50 mA) will be determined based on the comfort level of the patient after ensuring correct positioning. Correct positioning will be confirmed by observing a hallux reaction (plantar flexion of the big toe or, rarely, fanning of the fingers). T-MPNS sessions will be conducted twice a week for 6 weeks, with each session lasting 30 minutes. The intervention will consist of a 12-session T-MPNS treatment program.
  Interventions: Other: Transcutaneous medial plantar nerve stimulation (T-MPNS)
- Sham T-MPNS (Sham Comparator): In the Sham T-MPNS group, patients will receive stimulation with the same electrotherapy device, same patient and electrode positioning, and identical current characteristics as the T-MPNS group. Channel 2 of the device will be connected to the patient without delivering stimulation, while channel 1 will not be connected but will display current intensity and treatment duration on the device screen. The current intensity on channel 1 will only be able to be increased up to 2-3 mA to prevent patients from exceeding this level. Patients will be advised that higher stimulations might negatively affect treatment outcomes. All patients, including those in the placebo group, will be informed that the absence of motor or sensory responses during treatment does not imply ineffectiveness, alleviating concerns about lack of sensation. Sham T-MPNS sessions will be conducted twice weekly for 6 weeks, with each session lasting 30 minutes, totaling 12 sessions.
  Interventions: Other: Sham Transcutaneous medial plantar nerve stimulation (T-MPNS)

INTERVENTIONS:
Other: Transcutaneous medial plantar nerve stimulation (T-MPNS) — T-MPNS will be conducted unilaterally in the supine position using the electrotherapy device with surface electrodes. Two round self-adhesive electrodes will be positioned, with the negative electrode near the metatarsal-phalangeal joint of the great toe on the medial aspect of the foot and the positive electrode approximately 2 cm inferior-posterior to the medial malleolus (in front of the Medio-Malleolar-Calcaneal axis). Channel 1 will provide active stimulation, while channel 2 will remain inactive.
  Arms: T-MPNS
Other: Sham Transcutaneous medial plantar nerve stimulation (T-MPNS) — Sham T-MPNS group will be stimulated using the same electrotherapy device, with patients positioned identically and electrodes placed in the same positions as in the T-MPNS group. The current characteristics (pulse frequency 20 Hz and pulse width 200 ms) will also remain consistent across both channels. The second channel of the stimulation device will be designated as the channel connected to the patient but without delivering stimulation.
  Arms: Sham T-MPNS

SUMMARY:
The investigators conducted a prospective, randomized double-blind, placebo-controlled study based on a placebo technique to evaluate the efficacy of T-MPNS vs placebo in women with idiopathic OAB.

The main questions aimed to be answered are:

What are the effects of Transcutaneous Medial Plantar Nerve Stimulation (T-MPSS) on clinical parameters related to incontinence and quality of life compared to the placebo group in women with idiopathic overactive bladder (OAB)? Participants (n:40) with idiopathic OAB who meet the exclusion and inclusion criteria will be divided into 2 groups using a randomization table. The first group will receive T-MPSS (n:20) and the second group will receive placebo T-MPSS (n:20). Measurements will be performed twice in total, before and at the end of treatment (6th week).

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 with clinical diagnosis of idiopathic OAB
* Not tolerated or unresponsive to antimuscarinics and discontinued at least 4 weeks
* Able to understand the procedures, advantages and possible side effects
* Willing and able to complete the voiding diary and QoL questionnaire
* The strength of pelvic floor muscles 3/5 and more

Exclusion Criteria:

* Women with stress urinary incontinence
* History of conservative therapy (T-MPNS and Transcutaneous Tibial Nerve Stimulation/PTNS) within 6 months
* Pregnancy or intention to become pregnant during the study
* Current vulvovaginitis or urinary tract infections or malignancy
* Anatomic or posttraumatic malformations/skin disorders of medial plantar nerve region on inner foot that cannot allow to apply the electrodes
* More than stage 2 according to the pelvic organ prolapse quantification (POP-Q)
* Cardiac pacemaker, implanted defibrillator
* Previous urogynecological surgery within 3 months
* Neurogenic bladder, signs of neurologic abnormalities at objective examination; history of the peripheral or central neurologic pathology
* Ultrasonographic evidence of post-void residual volume more than 100 ml

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-11-28 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Improvement in incontinence episodes | Change from baseline Improvement in incontinence episodes at the 6th week after the treatment
  Reduction in incontinence episodes will be collected. Women with ≥50% reduction in incontinence episodes will be considered positive responders

SECONDARY OUTCOMES:
The severity of incontinence | Change from baseline the severity of incontinence at the 6th week after the treatment
  The 24-hour pad test was carried out to evaluate the severity of incontinence
Symptom severity | Change from baseline symptom severity at the 6th week after the treatment
  Overactive Bladder Questionnaire (OAB-V8) will be used to evaluate symptom severity in women with OAB in the study. The OAB-V8 consists of 8 questions in which patients can be classified as symptom severity: none (0), very little (1), a little (2), quite a few (3), very (4), and too many (5). The total score ranges from 0-40.
Frequency of voiding, nocturia, number of pads | Change from baseline Frequency of voiding, nocturia, number of pads at the 6th week after the treatment
  The frequency of voiding, nocturia, and the number of pads used will be collected from the 3-day bladder diary.
The Quality of Life | Change from baseline the Quality of Life at the 6th week after the treatment
  The Quality of Life-Incontinence Impact Questionnaire (IIQ7) will be used to assess specific QoL related to incontinence
Anxiety and Depression level | Change from baseline anxiety and Depression level at the 6th week after the treatment
  The Hospital Anxiety and Depression Scale (HAD), validated and reliability tested in Turkey in 1987, assesses levels of anxiety and depression. It comprises 14 questions, seven for anxiety and seven for depression, scored on a four-point Likert scale. Scores are summed for each subscale: questions 1, 3, 5, 7, 9, 11, and 13 for anxiety, and questions 2, 4, 6, 8, 10, 12, and 14 for depression. In Turkey, cutoff scores are 10/11 for anxiety and 7/8 for depression, indicating risk.
Assessment of sexual functions Assessment of sexual functions | Change from baseline assessment of sexual functions at the 6th week after the treatment
  In the evaluation of sexual function, the Female Sexual Function Index questionnaire is used, consisting of 19 questions assessing six main factors: sexual desire, arousal, lubrication, orgasm, satisfaction, and pain/discomfort. The highest possible total raw score is 95, while the lowest is 4. After multiplying the coefficients, the highest score is 36, and the lowest is 2. Impact coefficients used for scoring are: 0.6 for sexual desire, 0.3 for arousal and lubrication, and 0.4 for orgasm, satisfaction, and pain/discomfort. An Female Sexual Function Index score below 26.55 is indicative of sexual dysfunction
Cure and improvement rates | Change from baseline cure and improvement rates at the 6th week after the treatment
  Cure and improvement rates will be recorded in all groups at the end-of-treatment assessments. Values under 1.3 g in the 24-hour pad test will be considered as "cure", while a 50% or greater reduction in wet weight compared to baseline measurements at the end of treatment will be considered as "improvement".
Treatment Satisfaction Level | Change from baseline Treatment Satisfaction Level at the 6th week after the treatment
  At the end of the treatment, participants will be asked to evaluate their satisfaction level with the administered treatment using a Likert scale ranging from 1 to 5 (5=very satisfied, 4=satisfied, 3=neither satisfied nor dissatisfied, 2=dissatisfied, 1=very dissatisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Necmettin Yıldız, Prof., Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bo K, Frawley HC, Haylen BT, Abramov Y, Almeida FG, Berghmans B, Bortolini M, Dumoulin C, Gomes M, McClurg D, Meijlink J, Shelly E, Trabuco E, Walker C, Wells A. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for the conservative and nonpharmacological management of female pelvic floor dysfunction. Int Urogynecol J. 2017 Feb;28(2):191-213. doi: 10.1007/s00192-016-3123-4. Epub 2016 Dec 5. PMID 27921161
- [Background] C.K. Harding, M.C. Lapitan, S. Arlandis, K. Bø, H. Cobussen-Boekhorst, E. Costantini, et al. The European Association of Urology (EAU) Guidelines. EAU Guidelines on Management of Non-Neurogenic Female Lower Urinary Tract Symptoms. In: EAU Guidelines, 2023 (Internet). Available online at: https://uroweb.org/guidelines/non-neurogenic-female-luts
- [Background] Gormley EA, Lightner DJ, Faraday M, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline amendment. J Urol. 2015 May;193(5):1572-80. doi: 10.1016/j.juro.2015.01.087. Epub 2015 Jan 23. PMID 25623739
- [Background] de Groat WC, Yoshimura N. Anatomy and physiology of the lower urinary tract. Handb Clin Neurol. 2015;130:61-108. doi: 10.1016/B978-0-444-63247-0.00005-5. PMID 26003239
- [Background] de Groat WC, Griffiths D, Yoshimura N. Neural control of the lower urinary tract. Compr Physiol. 2015 Jan;5(1):327-96. doi: 10.1002/cphy.c130056. PMID 25589273
- [Background] Sonmez R, Yildiz N, Alkan H. Efficacy of percutaneous and transcutaneous tibial nerve stimulation in women with idiopathic overactive bladder: A prospective randomised controlled trial. Ann Phys Rehabil Med. 2022 Jan;65(1):101486. doi: 10.1016/j.rehab.2021.101486. Epub 2021 Nov 11. PMID 33429090
- [Background] Yildiz N, Sonmez R. Transcutaneous medial plantar nerve stimulation in women with idiopathic overactive bladder. Investig Clin Urol. 2023 Jul;64(4):395-403. doi: 10.4111/icu.20230009. PMID 37417565
- [Background] Burgio KL, Goode PS, Locher JL, Umlauf MG, Roth DL, Richter HE, Varner RE, Lloyd LK. Behavioral training with and without biofeedback in the treatment of urge incontinence in older women: a randomized controlled trial. JAMA. 2002 Nov 13;288(18):2293-9. doi: 10.1001/jama.288.18.2293. PMID 12425706
- [Background] Tezer T, Yildiz N, Sarsan A, Alkan H. Short-term effect of magnetic stimulation added to bladder training in women with idiopathic overactive bladder: A prospective randomized controlled trial. Neurourol Urodyn. 2022 Aug;41(6):1380-1389. doi: 10.1002/nau.24957. Epub 2022 May 20. PMID 35593007
- [Background] Yamanishi T, Homma Y, Nishizawa O, Yasuda K, Yokoyama O; SMN-X Study Group. Multicenter, randomized, sham-controlled study on the efficacy of magnetic stimulation for women with urgency urinary incontinence. Int J Urol. 2014 Apr;21(4):395-400. doi: 10.1111/iju.12289. Epub 2013 Oct 14. PMID 24118165
- [Background] Firinci S, Yildiz N, Alkan H, Aybek Z. Which combination is most effective in women with idiopathic overactive bladder, including bladder training, biofeedback, and electrical stimulation? A prospective randomized controlled trial. Neurourol Urodyn. 2020 Nov;39(8):2498-2508. doi: 10.1002/nau.24522. Epub 2020 Sep 22. PMID 32960999
- [Background] O'Sullivan R, Karantanis E, Stevermuer TL, Allen W, Moore KH. Definition of mild, moderate and severe incontinence on the 24-hour pad test. BJOG. 2004 Aug;111(8):859-62. doi: 10.1111/j.1471-0528.2004.00211.x. PMID 15270937
- [Background] Tarcan T, Mangır N, Özgür MÖ, Akbal C. OAB-V8 Overactive Bladder Questionnaire Validation Study. (Turkish) Üroloji Bülteni 2012;21:113-116. http://www.kontinansdernegi.org/userfiles/media/kontinans.galenos.com.tr/oab-v8-asiri-aktif-mesane-sorgulama-formu.pdf
- [Background] Acquadro C, Kopp Z, Coyne KS, Corcos J, Tubaro A, Choo MS, Oh SJ. Translating overactive bladder questionnaires in 14 languages. Urology. 2006 Mar;67(3):536-40. doi: 10.1016/j.urology.2005.09.035. PMID 16527574
- [Background] Cam C, Sakalli M, Ay P, Cam M, Karateke A. Validation of the short forms of the incontinence impact questionnaire (IIQ-7) and the urogenital distress inventory (UDI-6) in a Turkish population. Neurourol Urodyn. 2007;26(1):129-33. doi: 10.1002/nau.20292. PMID 17083117
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Aydemir Ö, Güvenir T, Küey L ve ark. (1987) Hastane Anksiyete ve Depresyon Ölçeği Türkçe Formunun Geçerlilik ve Güvenirliliği. Türk Psikiyatri Dergisi, 8:280-287
- [Background] Aygin, D., & Aslan, F. E. (2005). Kadin cinsel işlev ölçegi'nin Türkçeye uyarlamasi. Turkiye Klinikleri Journal of Medical Sciences, 25(3), 393-399
- [Background] Kim SJ, Choi HW, Cho HJ, Hwang TK, Kim JC. The influence of preoperative bladder outlet obstruction on continence and satisfaction in patients with stress urinary incontinence after midurethral sling. Int Neurourol J. 2010 Dec;14(4):267-71. doi: 10.5213/inj.2010.14.4.267. Epub 2010 Dec 31. PMID 21253340
- [Background] Finazzi-Agro E, Petta F, Sciobica F, Pasqualetti P, Musco S, Bove P. Percutaneous tibial nerve stimulation effects on detrusor overactivity incontinence are not due to a placebo effect: a randomized, double-blind, placebo controlled trial. J Urol. 2010 Nov;184(5):2001-6. doi: 10.1016/j.juro.2010.06.113. Epub 2010 Sep 20. PMID 20850833